CLINICAL TRIAL: NCT05149859
Title: Reconsidering Severity Classification for Binge Eating Disorder (BED): the Role of Impulsivity, Compulsivity and Co-occurring Disorders
Brief Title: Compuls-BED-Severity
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other); Centre d'expertise Poids, Image et Alimentation (CEPIA) (Unknown)
Responsible Party: Principal Investigator, Sylvain Iceta, Principal Investigator, Laval University
Other Study IDs: 2022-3743, 22144
Record Dates: First submitted 2021-11-19; First posted 2021-12-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Binge-Eating Disorder
Keywords: Binge-Eating Disorder; Impulsivity; Obesity; Attention; Emotional regulation
MeSH Terms: conditions — Binge-Eating Disorder; Impulsive Behavior; Obesity; Emotional Regulation | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- BED+ : Participants with obesity and binge eating disorder: Obesity is define by a BMI ≥ 30 kg.m-2 Binge eating disorder is defined by Binge Eating Disorder Screener (BEDS)-7 positive score and a Binge Eating Scale score >16
  Interventions: Other: Observational
- BED-: Participants with obesity but without binge eating disorder: Obesity is define by a BMI ≥ 30 kg.m-2 Binge eating disorder is defined by Binge Eating Disorder Screener (BEDS)-7 negative score and a Binge Eating Scale score < 12
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — (no intervention)

SUMMARY:
* Binge Eating Disorder (BED) has been fairly recently introduced into the Diagnostic and Statistical Manual 5 psychiatric classification and its severity criteria are still not well established.
* Moreover, it remains unclear whether BED is associated with greater metabolic severity or more somatic comorbidities, especially in obesity.
* Improved BED severity staging could lead to a better definition of management strategies and , therefore, facilitate screening and care.

The investigators' hypothesis is that an improved assessment of the impulsivity-compulsivity spectrum, emotional regulation, attentional impairment and somatic or psychiatric comorbidities will result in a better distinction between the severe form of BED (e.g., highly impulsive and somatically complicated) from milder form (e.g., more compulsive and less somatically complicated).

ELIGIBILITY:
Inclusion Criteria:

* men or women aged 1
* participants eligible for bariatric surgery (BMI>40, or BMI>35 with severe comorbidities)
* participants scheduled for medical evaluation and treatment of obesity at the IUCPQ Obesity Clinic (BMI≥30)
* participants scheduled for evaluation and treatment of BED at the CEPIA with obesity (BMI≥30)
* for the group with BED: positive BEDS-7 screen and Binge Eating Scale score >16;
* for the control group: have a negative BEDS-7 screen and Binge Eating Scale score<12
* be fluent in French and able to consent.

Exclusion criteria :

* participants with severe neurological disorder and/or major neurocognitive deficits;
* participants with previous bariatric surgery or with introduction or change of anti-obesity medication (liraglutide or naltrexone/bupropion) in the previous 3 months;
* participants who cannot read and/or understand French;
* participants under guardianship or curatorship;
* participants already included in a study with a conflict of interest with this study;
* inability to use a computer or iPad;
* inability to access an Internet connection or to visit one of the inclusion sites.

Secondary exclusion criteria:

* participants with a discordance between BEDS-7 (positive) and Binge Eating Scale (score ≤ 16) results found secondarily
* participants who did not participate in part of the assessments (e.g., self-questionnaires or neurocognitive tests) and participants with a rate of missing data>10%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from 2 sites: 1) the Institut Universitaire de Cardiologie et Pneumologie de Québec (IUCPQ; pre-bariatric surgery consultation and obesity care consultation); 2) the Centre d'Expertise Poids, Image et Alimentation (CEPIA), a clinic of the Institute of Nutrition and Functional Foods of Laval University (eatinig disorders consultation). The pre-selection of participants will be done using available data and screening tests deployed through the management frameworks already in place at the two sites. If needed, patients will be recruited by advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical and psychological comorbidities | Inclusion
  Number of current associated comorbidities to patient with and without BED
Binge Eating Scale score | Inclusion
  To assess binge eating severity based on the 16-item scale developed by Gormally et al in 1982

SECONDARY OUTCOMES:
Body Mass Index in kg.m-2 | Inclusion
  [Anthropometric markers] weight and height will be combined to report BMI in kg/m^2
Percentage of fat mass in % | Inclusion
  [Anthropometric markers] Based on impedance data, percentage fat mass will be reported when available
Waist and hip circumferences in cm | Inclusion
  [Anthropometric markers] Waist, hip circumference and Waist-hip ratio will be reported in cm when available
Triglycerides in mmol/L | Inclusion
  Routine clinical biological markers; part of lipidic profile (when available)
Cholesterol HDL and LDL in mmol/L | Inclusion
  Routine clinical biological markers; part of lipidic profile (when available)
Fasting blood glucose in mmol/L | Inclusion
  Routine clinical biological markers, when available.
Glycated hemoglobin (HbA1C) in % | Inclusion
  Routine clinical biological markers, when available.
Insulin in pmol/L | Inclusion
  Routine clinical biological markers, when available.
Visceral Adiposity Index | Inclusion
  The Visceral Adiposity Index (VAI) is a sex-specific mathematical index, based on Waist Circumference (WC), Body Mass Index (BMI), triglycerides (TG) and HDL cholesterol (HDL) levels, indirectly expressing visceral adipose function and insulin sensitivity.
UPPS-P Impulsive Behavior Scale short version, S-UPPS-P | Inclusion
  To assess the Impulsivity-compulsivity spectrum
Obsessive-Compulsive Inventory-Revised, OCI-R | Inclusion
  To assess the Impulsivity-compulsivity spectrum
Stop Signal Task | Inclusion
  To assess the Impulsivity-compulsivity spectrum
Difficulties in emotion regulation scale short form, DERS | Inclusion
  To assess the emotion regulation spectrum
Emotional Go / No-Go Task | Inclusion
  To assess the emotion regulation spectrum
Adult Attention Deficit Hyperactivity Disorder Self-Report Scale, ASRS | Inclusion
  To assess attentional functions
Integrated Visual and Auditory Continuous Performance Test, IVA-CPT | Inclusion
  To assess attentional functions
General Anxiety Disorder (GAD)-7 | Inclusion
  To assess anxiety disorders risk
Patient Health Questionnaire (PHQ)-9 | Inclusion
  To assess depression disorder risk

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Iceta, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (2):
- Canada (2):
  - Centre d'expertise Poids, Image et Alimentation (CEPIA), Québec
  - IUCPQ, Québec

IPD SHARING:
Plan to Share IPD: Undecided